CLINICAL TRIAL: NCT05853666
Title: Connecting Families to Improve Parental Self-efficacy and Parent Psychosocial and Infant Health Outcomes in the NICU Using an eHealth Solution (The CONNECT Study)
Brief Title: Connecting Families to Improve Parental Self-efficacy and Parent Psychosocial and Infant Health Outcomes in the NICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marsha Campbell-Yeo, Professor, Dalhousie University, School of Nursing, Faculty of Health, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CONNECT 1028664
Record Dates: First submitted 2023-03-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Self Efficacy; Infant Development; eHealth; Mental Health Wellness 1
Keywords: Neonatal; Parents; Families; eHealth; Implementation; Parent mental health; Infant outcomes; Parent presence

STUDY DESIGN:
Intervention Model Description: The CONNECT study is an unblinded multicentre stepped wedge cluster randomized controlled trial guided by a Hybrid-1 design examining the effectiveness and implementation of CNH+ compared to usual care (control) across four Canadian NICUs. All sites will begin in the control period (baseline). Every 5 months, one site will be randomized to CNH+ using a stepped wedge design allowing for 4 sites with 5 measurement steps.
Masking Description: Participants enrolled in the study will be allocated based on whether the NICU is in the control or intervention condition on their admission date. Blinding to the intervention at the participant level (i.e., standard care or CNH+) is not possible. Although an attention control website was considered, this was not implemented to ensure the findings are relevant against existing standard care (i.e., no eHealth component). Blinding is not possible at the unit level due to the shift in communication that will occur (e.g., virtual rounds). Blinding will occur during data analyses by using an external statistician not familiar with the group allocations. Examiners completing the 18-month neurodevelopment outcomes work at arm's length to the NICU with no or little knowledge of ongoing NICU studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group with Standard Care (No Intervention): Consenting families in the NICU during the baseline control period will receive standard care as it is already provided at each site. Data collection procedures will mirror intervention groups to ensure comparable control data.
- Intervention Group Receiving CNH+ (Experimental): Eligible consenting families (following enrollment) will be provided a secure login code and instructions to access the CNH+ educational modules and to send and receive virtual calls and text messages. Parents will be asked to use CNH+ during their entire NICU stay. To ensure equity, interested families without a personal device to access CNH+ will be offered a study-provided iPad for the duration of their infant's stay. Parents will have access to CNH+ while on the unit and 6 months post-discharge.
  Interventions: Behavioral: CNH+

INTERVENTIONS:
Behavioral: CNH+ — CNH+ is a bundled intervention targeting all four of Bandura's factors associated with improved self-efficacy (i.e., Mastery [evidence-based parent targeted education platform]; Vicarious Experience [observing other families similar to them succeeding in a task i.e., videos and photos]; Verbal Persuasion [in-person/virtual medical rounds and provision of social support]; and Physiological States [notifications and encouragement through mHealth text messaging, parent feedback, and tailored clinical care pathway]).
  Arms: Intervention Group Receiving CNH+

SUMMARY:
Preterm infants, 1 in 12 Canadian births, are at a significant increased risk of poor health outcomes, resulting in high healthcare burden. Parents of these infants report lower self-efficacy and worse mental health when compared to parents of term infants. There is an urgent need to use effective ways to improve parental self-efficacy and associated parent psychosocial and infant health outcomes. To improve parent and baby outcomes, the investigators will build on an existing eHealth solution to create Chez NICU Home+ (CNH+), which offers web-based, parent-targeted, interactive educational tools, virtual communication, and text message support during a baby's NICU stay. We will evaluate whether Chez NICU Home+ improves parental self-efficacy (primary outcome), parent psychosocial, and infant health outcomes in parents of babies requiring a NICU stay, and the implementation (ease and uptake) of Chez NICU Home+ in multiple sites. This study will be a multicentre implementation study, with a stepped wedge cluster randomized controlled trial across four Canadian NICUs. At the beginning of the study, data regarding current care will be collected from all sites to determine a baseline. Following baseline data collection, every five months one of the sites will start using the Chez NICU Home+ solution. A total of 800 parents and their babies, who are expected to stay at least 5 days in the NICU, will be recruited. Parents will complete a survey on psychosocial adjustment and infant outcomes when the study begins, as well as at 14 and 21 days after enrollment, at infant discharge from the NICU, and at 6 months post-discharge. Infant health and development outcomes will be collected at discharge, 6 and 18 months post-discharge via health records. The investigators predict that Chez NICU Home+ will be a positive, interactive care option, combining virtual parent education, tailored communication, and support, which will improve parental self-efficacy and parent psychosocial and infant health outcomes, and have long-term benefits for families.

ELIGIBILITY:
Inclusion Criteria:

* Parents who have an infant admitted to the NICU
* Parents who provide consent to participate within 7 days following birth
* Infant (regardless of gestational age or diagnosis) is anticipated to have at least a 5-day NICU stay

Exclusion Criteria:

* Parents who are unable to read or write English
* Parents whose infant is not anticipated to survive within the 7-day enrollment period after birth based on attending physician assessment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline parental self-perceived self-efficacy (as measured by the Perceived Maternal Parenting Self-Efficacy tool) at infant discharge date (immediately after the infant is discharged from the NICU) | At baseline and immediately after the infant is discharged from the NICU (the end of in-hospital phase)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental self-efficacy at their infant's discharge from the NICU? Measured using the Perceived Maternal Parenting Self-Efficacy (PMPS-E) tool at enrollment (baseline) and immediately after the discharge from the NICU of the infant admitted to the NICU, which marks the end of the in-hospital phase. All primary parent/caregiver(s) (up to 3) will be asked to complete this measure. The PMPS-E has a minimum score of 20 and a maximum score of 80. A higher score indicates a better outcome (higher levels of parental self-efficacy).
Change from baseline parental self-perceived self-efficacy (as measured by the Perceived Maternal Parenting Self-Efficacy tool) at 21 days (after the infant is born) | At baseline and 21 days after the infant is born
  In parents of NICU infants, does CNH+, when compared to standard care, change parental self-efficacy? Measured using the Perceived Maternal Parenting Self-Efficacy (PMPS-E) tool at enrollment (baseline) and 21 days after the infant admitted to the NICU is born. All primary parent/caregiver(s) (up to 3) will be asked to complete this measure. The PMPS-E has a minimum score of 20 and a maximum score of 80. A higher score indicates a better outcome (higher levels of parental self-efficacy).
Change from baseline parental self-perceived self-efficacy (as measured by the Perceived Maternal Parenting Self-Efficacy tool) at 6 months (after the infant is discharged from the NICU) | At baseline and 6 months after the infant is discharged from the NICU
  In parents of NICU infants, does CNH+, when compared to standard care, change parental self-efficacy 6 months after the infant is discharged from the NICU? Measured using the Perceived Maternal Parenting Self-Efficacy (PMPS-E) tool at enrollment, and 6 months after the infant is discharged from the NICU. All primary parent/caregiver(s) (up to 3) will be asked to complete this measure. The PMPS-E has a minimum score of 20 and a maximum score of 80. A higher score indicates a better outcome (higher levels of parental self-efficacy).

SECONDARY OUTCOMES:
Change from baseline parental level of stress (as measured using the State Trait Anxiety Inventory tool) at infant discharge date (immediately after the infant is discharged from the NICU) | At baseline and at infant discharge date (immediately after the infant is discharged from the NICU)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental level of stress at their infant's discharge from the NICU? Measured using the State Trait Anxiety Inventory (STAI) tool at enrollment (baseline) and immediately after the discharge from the NICU of the infant admitted to the NICU, which marks the end of the in-hospital phase. The primary parent/caregiver(s) will be asked to complete this measure. The STAI has a minimum score of 20 and a maximum score of 80. A higher score indicates a worse outcome (higher levels of parental anxiety).
Change from baseline parental level of stress (as measured using the State Trait Anxiety Inventory tool) at 21 days (after the infant is born) | At baseline and at 21 days (after the infant is born)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental level of stress at 21 days after the infant is born? Measured using the State Trait Anxiety Inventory (STAI) tool at enrollment (baseline) and at 21 days after the infant admitted to the NICU is born. The primary parent/caregiver(s) will be asked to complete this measure. The STAI has a minimum score of 20 and a maximum score of 80. A higher score indicates a worse outcome (higher levels of parental anxiety).
Change from baseline parental level of NICU-specific stressors (as measured using the Parental Stressor Scale tool) at infant discharge date (immediately after the infant is discharged from the NICU) | At baseline and at infant discharge date (immediately after the infant is discharged from the NICU)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental level of NICU-specific stressors at their infant's discharge from the NICU? Measured using the Parental Stressor Scale (PSS NICU) tool at enrollment (baseline) and immediately after the discharge from the NICU of the infant admitted to the NICU, which marks the end of the in-hospital phase. The primary parent/caregiver(s) will be asked to complete this measure. The PSS NICU has a minimum score of 18 and a maximum score of 90. A lower score indicates a better outcome (lower levels of parental NICU-specific stress).
Change from baseline parental level of NICU-specific stressors (as measured using the Parental Stressor Scale tool) at 21 days (after the infant is born) | At baseline and at 21 days (after the infant is born)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental level of NICU-specific stressors at 21 days after the infant is born? Measured using the Parental Stressor Scale (PSS NICU) tool at enrollment (baseline) and at 21 days after the infant admitted to the NICU is born. The primary parent/caregiver(s) will be asked to complete this measure. The PSS NICU has a minimum score of 18 and a maximum score of 90. A lower score indicates a better outcome (lower levels of parental NICU-specific stress).
Change from baseline parental level of depression (as measured using the Postpartum Depression Screening Scale tool) at infant discharge date (immediately after the infant is discharged from the NICU) | At baseline and at infant discharge date (immediately after the infant is discharged from the NICU)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental level of depression at their infant's discharge from the NICU? Measured using the Postpartum Depression Screening Scale (PDSS) tool at enrollment (baseline) and immediately after the discharge from the NICU of the infant admitted to the NICU, which marks the end of the in-hospital phase. The primary parent/caregiver(s) will be asked to complete this measure. The PDSS has a minimum score of 35 and a maximum score of 175. A higher score indicates a worse outcome (higher levels of postpartum depression).
Change from baseline parental level of depression (as measured using the Postpartum Depression Screening Scale tool) at 14 days (after the infant is born) | At baseline and at 14 days (after the infant is born)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental level depression at 14 days after the infant is born? Measured using the Postpartum Depression Screening Scale (PDSS) tool at enrollment (baseline) and at 14 days after the infant admitted to the NICU is born. The primary parent/caregiver(s) will be asked to complete this measure. The PDSS has a minimum score of 35 and a maximum score of 175. A higher score indicates a worse outcome (higher levels of postpartum depression).
Change from baseline parental level of depression (as measured using the Postpartum Depression Screening Scale tool) at 21 days (after the infant is born) | At baseline and at 21 days (after the infant is born)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental level depression at 21 days after the infant is born? Measured using the Postpartum Depression Screening Scale (PDSS) tool at enrollment (baseline) and at 21 days after the infant admitted to the NICU is born. The primary parent/caregiver(s) will be asked to complete this measure. The PDSS has a minimum score of 35 and a maximum score of 175. A higher score indicates a worse outcome (higher levels of postpartum depression).
Change from baseline parental quality of life (as measured using the Quality of Life (EQ-5D-5L) tool) at infant discharge date (immediately after the infant is discharged from the NICU) | At baseline and at infant discharge date (immediately after the infant is discharged from the NICU)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental quality of life at their infant's discharge from the NICU? Measured using the Quality of Life (EQ-5D-5L) tool at enrollment (baseline) and immediately after the discharge from the NICU of the infant admitted to the NICU, which marks the end of the in-hospital phase. The primary parent/caregiver(s) will be asked to complete this measure. The Quality of Life (EQ-5D-5L) has a descriptive score and a visual analog scale. The descriptive score has a minimum score of 5 and a maximum score of 25. A higher score indicates a worse outcome (lower levels of quality of life). The visual analog score has a minimum score of 0 and a maximum score of 100. A higher score indicates a better outcome (higher levels of quality of life).
Change from baseline parental quality of life (as measured using the Quality of Life (EQ-5D-5L) tool) at 21 days (after the infant is born) | At baseline and at 21 days (after the infant is born)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental quality of life at 21 days after the infant is born? Measured using the Quality of Life (EQ-5D-5L) tool at enrollment (baseline) and at 21 days after the infant admitted to the NICU is born. The primary parent/caregiver(s) will be asked to complete this measure. The Quality of Life (EQ-5D-5L) has a descriptive score and a visual analog scale. The descriptive score has a minimum score of 5 and a maximum score of 25. A higher score indicates a worse outcome (lower levels of quality of life). The visual analog score has a minimum score of 0 and a maximum score of 100. A higher score indicates a better outcome (higher levels of quality of life).
Perceived amount of family-centred care in the NICU (as measured using the Family Centred Care Scale tool) at infant discharge date (immediately after the infant is discharged from the NICU) | At infant discharge date (immediately after the infant is discharged from the NICU)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental perceived amount of family-centred care in the NICU at their infant's discharge from the NICU? Measured using the Family Centred Care Scale tool immediately after the discharge from the NICU of the infant admitted to the NICU. The primary parent/caregiver(s) will be asked to complete this measure. The Family Centred Care Scale has a minimum score of 20 and a maximum score of 80. A higher score indicates a better outcome (higher levels of perceived amount of family-centred care in the NICU).
Perceived amount of family engagement in care in the NICU (as measured using the CO-PARTNER Tool) at infant discharge date (immediately after the infant is discharged from the NICU) | At infant discharge date (immediately after the infant is discharged from the NICU)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental perceived amount of family engagement in care in the NICU at their infant's discharge from the NICU? Measured using the CO-PARTNER Tool immediately after the discharge from the NICU of the infant admitted to the NICU. The primary parent/caregiver(s) will be asked to complete this measure. The CO-PARTNER Tool has a minimum score of 0 and a maximum score of 62. A higher score indicates a better outcome (higher levels of positive inherent relationship between participation and collaboration).
Perceived parental readiness to have their infant discharged from the NICU and sent home (as measured using the Readiness for Hospital Discharge tool) at infant discharge date (immediately after the infant is discharged from the NICU) | At infant discharge date (immediately after the infant is discharged from the NICU)
  In parents of NICU infants, does CNH+, when compared to standard care, change parental perceived readiness to have their infant discharged from the NICU and sent home, at the time of their infant's discharge from the NICU? Measured using the Readiness for Hospital Discharge tool immediately after the discharge from the NICU of the infant admitted to the NICU. The primary parent/caregiver(s) will be asked to complete this measure. The Readiness for Hospital Discharge tool has a minimum average score of 0 and a maximum score of 10. A higher score indicates a better outcome (higher levels of readiness for hospital discharge).
Infant weight growth (change in weight since birth) at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change infant weight growth (change in weight since birth) at the infant's discharge from the NICU? Data collected by chart review.
Infant head growth (change in head circumference since birth) at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change infant head growth (change in head circumference since birth) at the infant's discharge from the NICU? Data collected by chart review.
Infant length of stay in the NICU (in days) at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change infant length of stay in the NICU (in days) at the infant's discharge from the NICU? Data collected by chart review.
Amount of provision of mothers' own breast milk for their infant during their infant's stay in the NICU, totalled at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In parents of NICU infants, does CNH+, when compared to standard care, change the amount of provision of mothers' own breast milk for their infant during their infant's stay in the NICU? Data collected by chart review.
Infant receipt of breast milk at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In parents of NICU infants, does CNH+, when compared to standard care, change the receipt of breast milk for their infant at the infant's discharge from the NICU? Data collected by chart review.
Amount of time for the infant to reach full enteral feeds during their stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the amount of time for the infant to reach full enteral feeds during their stay in the NICU? Data collected by chart review.
Incidence of mortality during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the incidence of mortality during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Incidence of necrotizing enterocolitis (Stage >II) during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the incidence of necrotizing enterocolitis (Stage >II) during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Incidence of late-onset sepsis during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the incidence of late-onset sepsis during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Incidence of chronic lung disease during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the incidence of chronic lung disease during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Incidence of retinopathy of prematurity (Stage ≥3) during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the incidence of retinopathy of prematurity (Stage ≥3) during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Incidence of severe brain injury during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the incidence of severe brain injury during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Incidence of treated Patent Ductus Arteriosus (PDA) during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the incidence of treated Patent Ductus Arteriosus (PDA) during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Incidence of air leak during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the incidence of air leak during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Duration of respiratory support (invasive and non-invasive) during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the duration of respiratory support (invasive and non-invasive) during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Duration of oxygen supplementation during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the duration of oxygen supplementation during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Duration of total parenteral nutrition (TPN) during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the duration of total parenteral nutrition (TPN) during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Duration of hypoxic ischemic encephalopathy (HIE) during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the duration of hypoxic ischemic encephalopathy (HIE) during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Number of infant's days with a central venous line in situ during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the number of infant's days with a central venous line in situ during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Number of infant central line-associated bloodstream infections during the infant's stay in the NICU, recorded at infant discharge date (immediately after the infant is discharged from the NICU). | At infant discharge date (immediately after the infant is discharged from the NICU)
  In NICU infants, does CNH+, when compared to standard care, change the number of infant central line-associated bloodstream infections during their stay in the NICU? Data are collected routinely via the Canadian Neonatal Network and abstracted for study use.
Infant neurological examination score at 18 months corrected gestational age | At 18 months of the infants corrected gestational age
  In NICU infants, does CNH+, when compared to standard care, improve infant neurodevelopment as measured through a neurological examination? Data are measured and collected at routine follow-up in NICUs at 18 months corrected gestational age.
Infant hearing assessment score at 18 months corrected gestational age | At 18 months of the infants corrected gestational age
  In NICU infants, does CNH+, when compared to standard care, improve infant neurodevelopment as measured through a hearing assessment? Data are measured and collected at routine follow-up in NICUs at 18 months corrected gestational age.
Infant vision assessment score at 18 months corrected gestational age | At 18 months of the infants corrected gestational age
  In NICU infants, does CNH+, when compared to standard care, improve infant neurodevelopment as measured through a vision assessment? Data are measured and collected at routine follow-up in NICUs at 18 months corrected gestational age.
Infant development score at 18 months corrected gestational age | At 18 months of the infants corrected gestational age
  In NICU infants, does CNH+, when compared to standard care, improve infant neurodevelopment as measured through the Bayley Scales of Infant and Toddler Development? Data are measured and collected at routine follow-up in NICUs at 18 months corrected gestational age.
Number of Chez NICU Home educational modules completed at 6 months after the discharge of the infant from the NICU. | At 6 months after the discharge of the infant from the NICU
  What number of Chez NICU Home educational modules are completed by parents of infants in the NICU at 6 months after the discharge of the infant from the NICU? Metrics data will be captured by the CNH platform.
Number of Chez NICU Home educational modules viewed at 6 months after the discharge of the infant from the NICU. | At 6 months after the discharge of the infant from the NICU
  What number of Chez NICU Home educational modules are viewed by parents of infants in the NICU at 6 months after the discharge of the infant from the NICU? Metrics data will be captured by the CNH platform.
Amount of time spent on the Chez NICU Home platform at 6 months after the discharge of the infant from the NICU. | At 6 months after the discharge of the infant from the NICU
  What amount of time do parents of infants in the NICU spend on the Chez NICU Home platform, at 6 months after the discharge of the infant from the NICU? Metrics data will be captured by the CNH platform.
Number of text messages received by parents of infants in the NICU, completed at 6 months after the discharge of the infant from the NICU. | At 6 months after the discharge of the infant from the NICU
  What number of text messages are received by parents of infants in the NICU at 6 months after the discharge of the infant from the NICU? Metrics data will be captured by TextIt application.
Number of virtual communication tools used by parents of infants in the NICU, completed at 6 months after the discharge of the infant from the NICU. | At 6 months after the discharge of the infant from the NICU
  What number of virtual communication tools are used by parents of infants in the NICU at 6 months after the discharge of the infant from the NICU? Metrics data will be captured by CNH+.
Number of parents of infants in the NICU who enroll in CNH+ when offered? | At baseline (upon enrollment to the study)
  What number of parents of infants in the NICU who enroll in CNH+ when offered at the beginning of the study?
Parents' perceived ease of use of the CNH+ intervention (as measured using the e-Health impact questionnaire) at 6 months after the discharge of the infant from the NICU) | At 6 months after the discharge of the infant from the NICU
  In parents of NICU infants, what are parents' perceived ease of use of the CNH+ intervention at 6 months after the discharge of the infant from the NICU)? Measured using the e-Health impact questionnaire tool 6 months after the discharge of the infant from the NICU. The primary parent/caregiver(s) will be asked to complete this measure. When scored, the e-Health impact questionnaire tool has a minimum score of 0 and a maximum score of 100. A higher score indicates a better outcome (higher levels of perceived ease of use).

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Campbell-Yeo, RN NNP PhD, Principal Investigator — Dalhousie University

IPD SHARING:
Plan to Share IPD: No